CLINICAL TRIAL: NCT05420220
Title: An Open-Label, Multi-Center, Phase 2 Clinical Study to Evaluate Efficacy, Safety, and Tolerability of KN046 in Combination With Axitinib in Subjects With Advanced Non-Small Cell Lung Cancer
Brief Title: Study of KN046 in Subjects With Advanced Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KN046-209
Record Dates: First submitted 2022-06-12; First posted 2022-06-15 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Advanced Non-small Cell Lung Cancer
MeSH Terms: interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KN046+Axitinib (Experimental): Eligible subjects will receive KN046 5 mg/kg Q3W IV in combination with Axitinib 5 mg bid po, until progressive disease as judged by the investigator per RECIST v1.1
  Interventions: Biological: KN046 (Recombinant Humanized PD-L1/CTLA-4 Bispecific Single Domain Antibody Fc Fusion Protein Injection); Combination Product: Axitinib

INTERVENTIONS:
Biological: KN046 (Recombinant Humanized PD-L1/CTLA-4 Bispecific Single Domain Antibody Fc Fusion Protein Injection) — 5 mg/kg Q3W IV
Combination Product: Axitinib — 5mg bid po

SUMMARY:
This is an open-label, multi-center, Phase 2 study in subjects with treatment-naïve locally advanced (unresectable and unable to receive radical chemoradiotherapy) or metastatic PD-L1-positive non-small cell lung cancer (NSCLC) who have received systemic therapy.

DETAILED DESCRIPTION:
Subjects should provide tumor sample slides at screening, and the central laboratory will confirm whether the PD-L1 expression meets the inclusion criteria. Eligible subjects will receive KN046 5 mg/kg Q3W IV in combination with Axitinib 5 mg bid po, until progressive disease as judged by the investigator per RECIST v1.1, clinical progression, unacceptable toxicity, 35 doses of KN046 treatment, initiation of new systemic anti-tumor therapy, death, loss to follow-up, voluntary withdrawal, or end of the study, whichever occurs first. Subjects who discontinue one of the two trial treatments (KN046 or Axitinib) for reasons other than progressive disease may continue monotherapy with the other trial treatment. From the date of the first dose, up to 35 doses of KN046 will be administered and Axitinib will be administered until progressive disease or intolerable toxicity. Treatment with KN046 may be modified by dose interruption. Treatment with Axitinib may be modified by dose interruption or dose reduction.

The screening period will last 28 days prior to the first dose. Subjects will undergo tumor assessments at screening, every 6 weeks (± 7 days) within 54 weeks after the first dose, and every 9 weeks (± 7 days) thereafter until progressive disease as judged by the investigator per RECIST v1.1, initiation of new systemic anti-tumor therapy, death, loss to follow-up, voluntary withdrawal, or end of the study, whichever occurs first. The investigator may decide whether to confirm the progressive disease at approximately 4 to 6 weeks (not earlier than 4 weeks and not later than 6 weeks) based on the clinical symptoms of the subject after the subject first develops radiographic progressive disease (PD) per RECIST v1.1. Prior to confirmation of the progressive disease, if the subject is clinically stable, the subject is allowed to continue to receive the study drug after discussion with the medical monitor and documentation until the investigator confirms that the subject is no longer benefiting from the study drug (up to 35 doses of KN046).

Subjects will have an end of treatment (EOT) visit within 7 days at the end of trial treatment regimen KN046/Axitinib (whichever occurs later), and a safety follow-up visit 30 days (± 7 days) after the last dose of KN046/Axitinib (whichever occurs later) or decision made to discontinue all trial treatments. A safety follow-up visit will be scheduled 90 days (± 14 days) after the last dose of KN046. For subjects who discontinue treatment with KN046 first and continue treatment with Axitinib, the safety follow-up visit 90 days after the last dose of KN046 is not required if 30 days after the last dose of Axitinib is later than 90 days after the last dose of KN046.

The information of survival status and subsequent anti-tumor therapy will be collected every 12 weeks (± 14 days) after the end of treatment. Survival follow-up will continue until the end of the study. The end of the study is defined as 1 year after the last dose of all subjects, or the completion of the last study-related telephone contact or visit of the last subject, withdrawal from the study or loss to follow-up (i.e., the investigator is unable to contact the subject), or death or premature withdrawal from the study of all subjects, or the sponsor assesses that the study has met the study expectations (e.g., completion of the primary endpoint assessments), whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* I01. Subjects who are able to understand the Informed Consent Form (ICF) and sign the ICF;
* I02. Male or female subjects, aged 18 years or older; willing and able to complete all required study procedures;
* I03. Subjects with histologically or cytologically confirmed locally advanced (stage IIIB/IIIC) and stage IV (defined by the Union for International Cancer Control and the American Joint Committee on Cancer Staging System, edition 8) non-small cell lung cancer that is unresectable and unable to receive radical chemoradiotherapy;
* I04. Subjects who are PD-L1+ (TPS ≥ 1%) confirmed by central laboratory;
* I05. Subjects who must have negative EGFR mutation and ALK translocation (testing is not mandatory for subjects with squamous cell carcinoma whose EGFR/ALK gene mutation status is unknown). Subjects with known driver genes for other approved targeted drug therapies are also not eligible.
* I06. Subjects who have not received systemic therapy for locally advanced/metastatic NSCLC. Subjects who have received prior neoadjuvant, adjuvant chemotherapy, or radical chemoradiotherapy are allowed if they develop progressive disease at least 6 months after completing the aforementioned treatment;
* I07. Subjects with at least one measurable lesion per RECIST v1.1 at baseline;
* I08. Subjects with a ECOG score of 0 or 1;
* I09. Subjects with adequate organ function assessed within 7 days prior to first trial treatment as follows:

  • Hematology (without transfusion or use of hematopoietic stimulators within 14 days prior to enrollment)
* ANC≥1.5 × 109/L;
* Hemoglobin ≥ 9 g/dL;
* Platelets ≥ 100 × 109/L;
* White blood cell count (WBC) ≥ 4.0 × 109/L and ≤ 15 × 109/L;

  • Renal function
* Serum creatinine ≤ 1.5 × upper limit of normal (ULN) or creatinine clearance ≥ 60 mL/min (calculated according to the Cockcroft-Gault method, see Appendix 7 for details);
* Urine protein < 2+ by urinalysis. If urine protein is ≥ 2+, the subject is eligible only if 24-hour urine protein is < 1.0 g/24 hours;

  • Hepatic function
* Total bilirubin ≤ 1.5 × ULN (≤ 3 × ULN for subjects with Giltert's syndrome);
* ALT/AST ≤ 2.5 × ULN (≤ 5.0 × ULN for subjects with liver metastases);

  • Coagulation
* INR or PT ≤ 1.5 × ULN
* aPTT≤1.5 × ULN;
* I10. Subjects with a left ventricular ejection fraction (LVEF) of ≥ 50% (by ECHO or MUGA assessment)
* I11. Subjects who have a life expectancy of ≥ 3 months;
* I12. Female subjects of childbearing potential who have a negative serum pregnancy test within 7 days prior to the first dose;

Exclusion Criteria

* E01. Subjects with untreated metastases to central nervous system. Subjects with a previous diagnosis of metastases to central nervous system are eligible to enroll if they have completed treatment, have been clinically stable (assessed by imaging, preferably MRI with contrast-enhanced MRI or CT) for at least 2 weeks, and their neurological and other clinical symptoms have recovered to ≤ Grade 1 per NCI-CTC AE at least 2 weeks before the first dose, and steroids for brain metastases are discontinued 7 days prior to the first dose of trial treatment.
* E02. Subjects who have received prior immune checkpoint inhibitors, including but not limited to anti-PD-1, PD-L1, CTLA-4, LAG3 agent or other immune checkpoint inhibitors; Subjects who have received prior treatment with single/multi-target inhibitors or monoclonal antibodies to VEGF or VEGFR signaling pathways;
* E03. Subjects who have undergone major surgery for any reason within 4 weeks prior to the first dose of trial treatment;
* E04. Subjects who have a history of radiotherapy that meets the following criteria and fail to recover from toxicity/complications of radiotherapy to ≤ Grade 1 per NCI-CTCAE (except alopecia and fatigue)

  1. Thoracic radiotherapy: subjects who have received a chest radiation dose of > 30 Gy within 24 weeks before the first dose;
  2. Non-thoracic radiotherapy: subjects who have received a non-thoracic radiotherapy with a dose of > 30 Gy within 4 weeks before the first dose.
  3. Subjects who have received palliative radiotherapy with a dose of ≤ 30 Gy within 2 weeks before the first dose; Palliative radiotherapy for symptom control is permitted and must be completed at least 2 weeks before the start of study drug.
* E05. Subjects who have participated in a study or received the treatment with other investigational drugs within 4 weeks or less than 5 times of half-life (not less than 2 weeks), whichever is shorter prior to the first dose of trial treatment;
* E06. Subjects who have received treatment with anti-tumor vaccines, anti-tumor traditional Chinese medicine or other anti-tumor drugs with immunostimulatory effects within 2 weeks prior to the first dose;
* E07. Subjects who require systemic corticosteroids (≥ 10 mg/day prednisone or equivalent dose of other corticosteroids) or immunosuppressive therapy for 7 consecutive days within 14 days prior to the first dose; except inhaled or topical corticosteroids, or physiologic replacement doses of corticosteroids for adrenal insufficiency; short-term (≤ 7 days) corticosteroids are allowed for prophylaxis (e.g., contrast media allergy) or for the treatment of non-autoimmune disorders (e.g., delayed-type hypersensitivity reactions due to contact allergens);
* E08. Subjects who have received vaccination within 28 days prior to the first dose of trial treatment, except for inactivated vaccines.
* E09. Subjects who have interstitial lung disease, or a history of pneumonia requiring oral or intravenous corticosteroids to assist in management;
* E10. Subjects with uncontrolled hypertension (blood pressure ≥ 150/95 mmHg at rest) after standard antihypertensive therapy.
* E11. Subjects who have a history of or current autoimmune diseases, including, but not limited to, Crohn's disease, ulcerative colitis, systemic lupus erythematosus, sarcoidosis, Wegener's syndrome (granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis), autoimmune hepatitis, systemic sclerosis (scleroderma, etc.), Hashimoto's thyroiditis (refer to the following exceptions), autoimmune vasculitis, autoimmune neuropathy (Guillain-Barre syndrome).
* E12. Subjects who have other malignancies within 5 years before the first dose, except cured skin squamous cell carcinoma, basal cell carcinoma, non-muscle invasive bladder cancer, localized low-risk prostate cancer (defined as stage ≤ T2a, Gleason score ≤ 6, and PSA ≤ 10 ng/mL (as measured) at diagnosis of prostate cancer, the subjects had received curative treatment and no prostate-specific antigen (PSA) biochemical recurrence), and in-situ cervical/breast cancer;
* E13. Subjects with uncontrolled comorbidities, including but not limited to:

  * Active HBV or HCV infection;
  * Known HIV infection or known history of acquired immune deficiency syndrome (AIDS);
  * Active tuberculosis infection;
  * Active infection within 4 weeks prior to the first dose of trial treatment that requires the use of systemic antibiotics ≥ 7 days;
  * Subjects with uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated (monthly or more frequent) drainage
  * Clinically significant (that is, active) cardiovascular disease:
  * Uncontrolled ≥ Grade 3 active hemorrhage by medical intervention within 4 weeks prior to the first dose of trial treatment;
  * Subjects who require long-term anticoagulant therapy with warfarin (prophylactic anticoagulation for maintenance of the venous access device is permitted); Subjects who require long-term antiplatelet therapy (e.g., aspirin or clopidogrel at loading dose; or aspirin at maintenance dose of ≥ 100 mg/day; or clopidogrel at maintenance dose of ≥ 75 mg/day).
  * Serious, non-healing wound, ulcer, or bone fracture;
* E14. Subjects whose tumor has invaded important blood vessels or, as judged by the investigator, the tumor is highly likely to invade important blood vessels and cause major hemorrhage during treatment.
* E15. Subjects with impaired gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of Axitinib, including but not limited to:

  * Inability to take oral medication
  * Prior surgical procedures affecting absorption including total/partial gastric resection;
  * Malabsorption syndromes, uncontrolled nausea, vomiting, diarrhea.
* E16. Subjects with current use or anticipated need for treatment with drugs or foods that are known strong CYP3A4/5 inhibitors or CYP3A4/5 inducers within 14 days prior to the first dose of trial treatment (e.g., grapefruit juice or grapefruit/grapefruit-related citrus fruits [e.g., oranges, pomelos], ketoconazole, miconazole etc. ). The topical use of these medications (if applicable) such as 2% ketoconazole cream is allowed;
* E17. Subjects with current use or anticipated need for treatment with drugs that are known strong CYP3A4/5 inducers within 14 days prior to enrollment or thereafter (e.g., phenobarbital, rifampin);
* E18. Subjects with toxicity related to prior therapy (including any prior investigational therapy) that has not recovered to ≤ Grade 1 per CTCAE (NCI-CTCAE v5.0) or baseline, except for alopecia of any grade;
* E19. Subjects who have received prior allogeneic hematopoietic stem cell transplantation or solid organ transplantation;
* E20. Subjects who have known serious hypersensitivity to antibody drugs (≥ Grade 3 per NCI-CTCAE v5.0), any history of serious drug hypersensitivity (e.g., immune-mediated hepatotoxicity, immune-mediated thrombocytopenia or anemia); or known allergy to the study drug or any of its excipients
* E21. Pregnant or lactating women;
* E22. Subjects with other medical conditions that at the discretion of investigator affect the safety or efficacy assessment or treatment compliance of the trial. These include, but are not limited to, mental illness, alcoholism, drug addiction or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2027-05-29 (Estimated); Study Completion 2027-12-26 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  defined as the proportion of subjects with a confirmed best overall response (BOR) of CR or PR per RECIST v1.1 as assessed by the investigator.

SECONDARY OUTCOMES:
Duration of response (DOR) | Up to 2 years
  defined as the time from the first documentation of CR or PR to the first documentation of progressive disease or death due to any cause (whichever occurs first);
Disease control rate (DCR) | Up to 2 years
  defined as the proportion of subjects with a best overall response of CR, PR or SD;
Clinical benefit rate (CBR), | Up to 2 years
  defined as the proportion of subjects with a best overall response of CR, PR, or SD ≥ 24 weeks;
Time to response (TTR) | Up to 2 years
  defined as the time from the first trial treatment to the first documentation of objective response (CR or PR);
Progression-free survival (PFS) | Up to 2 years
  defined as the time from the first trial treatment to progressive disease or death due to any cause (whichever occurs first);
Overall survival (OS) | Up to 2 years
  defined as the time from the first trial treatment to death due to any cause.
Incidence and severity (as graded by CTCAE v5.0) of treatment-emergent adverse events (TEAEs), | Up to 2 years
  Incidence and severity (as graded by CTCAE v5.0) of treatment-emergent adverse events (TEAEs), abnormal laboratory values, and abnormal physical examinations.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Doctor, Principal Investigator — Sun Yat-sen University
Locations (6):
- China (6):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - The first affiliated hospital, Zhejiang university, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No